CLINICAL TRIAL: NCT01123928
Title: The Effect of Counseling in Cataract Screening: Guangdong Uptake of Surgery Trial
Brief Title: Guangdong Uptake of Surgery Trial
Acronym: GUSTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Swarthmore College (Other); Helen Keller International (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Dr. Nathan Congdon, MD, MPH, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZOC-123
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Results first posted 2012-02-02 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Cataract
Keywords: cataract; counseling; surgical uptake; follow-up
MeSH Terms: conditions — Cataract | interventions — Videotape Recording; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling (Experimental): Subjects will be asked to watch a 5-10 min video and participate in a 10-15 min pre-operative counseling session with a trained nurse. Subjects will also participate in a 5 min post-operative counseling session.
  Interventions: Behavioral: Video and counseling for cataract patients
- Non-counseling (No Intervention)

INTERVENTIONS:
Behavioral: Video and counseling for cataract patients — Intervention includes: (1) a 5-10 min video consisting of testimony from a previous cataract patient and a doctor; (2) a 10-15 min pre-operative counseling session with a trained nurse, and (3) a 5 min post-operative counseling session with a trained nurse.
  Arms: Counseling

SUMMARY:
The purpose of this study is:

1. To determine whether an educational intervention designed based on studies in the area is effective in increasing acceptance of surgery and presentation to the hospital, when adjusting for a number of potential determinants of service uptake;
2. To assess short-term impact of the educational intervention on knowledge about cataract and attitudes toward locally-available surgical services.

DETAILED DESCRIPTION:
China is home to the 18% of the world's blind people, an estimated 6.6 million. In China, cataract is the leading cause of blindness. In Guangdong, current counseling measures for patients diagnosed with cataract are minimal and often lack adequate descriptions of what cataract is, what causes cataract, and benefits/risks of surgery. A counseling session for cataract patients and family members, conducted by a trained nurse during outreach screening, may increase subsequent attendance at pre-operative examination, acceptance of cataract surgery, and attendance at follow-up examinations. An integral part of this counseling is a short movie consisting of testimony from a former cataract patient who underwent surgery ("pseudophakic motivator"). The use of pseudophakic motivators have been shown to be effective in increasing surgical uptake. In addition, a previously validated "Barriers Questionnaire" will be used to assess predictors of of hospital attendance, surgery acceptance, and follow-up attendance in the categories of cost, transportation, knowledge, and concerns about quality.

ELIGIBILITY:
Inclusion Criteria:

* thought by the examiner to have age-related or myopic cataract in one or both eyes
* pinhole-corrected visual acuity less than or equal to 6/18.

Exclusion Criteria:

* traumatic cataract
* inability to give informed consent due to dementia or other reasons.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Mingguang He, PHD, MPH, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; David Friedman, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Tan L. Increasing the volume of cataract surgery: an experience in rural China. Community Eye Health. 2006 Dec;19(60):61-3. No abstract available. PMID 17515966
- [Background] Ellwein LB, Lepkowski JM, Thulasiraj RD, Brilliant GE. The cost effectiveness of strategies to reduce barriers to cataract surgery. The Operations Research Group. Int Ophthalmol. 1991 May;15(3):175-83. doi: 10.1007/BF00153924. PMID 1904845
- [Derived] Liu T, Congdon N, Yan X, Jin L, Wu Y, Friedman D, He M. A randomized, controlled trial of an intervention promoting cataract surgery acceptance in rural China: the Guangzhou Uptake of Surgery Trial (GUSTO). Invest Ophthalmol Vis Sci. 2012 Aug 13;53(9):5271-8. doi: 10.1167/iovs.12-9798. PMID 22789919
- [Derived] Barry MP, Dagnelie G; Argus II Study Group. Use of the Argus II retinal prosthesis to improve visual guidance of fine hand movements. Invest Ophthalmol Vis Sci. 2012 Aug 1;53(9):5095-101. doi: 10.1167/iovs.12-9536. PMID 22661464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 32 outreach screening sessions in various villages and townships of Guangdong province from June 2010 to November 2010.
Groups:
- Non-counseling: Subjects will be told that they had decreased vision due to cataract and that this could be treated, without being shown the video or given the counseling session by the nurse.
Period: Overall Study
Arm/Group | Counseling | Non-counseling
Started | 212 | 222
Completed | 212 | 222
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counseling | Non-counseling | Total
Number analyzed (Participants) | 212 | 222 | 434
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 19 | 48
  >=65 years | 183 | 203 | 386
Age Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8.7) | 75.5 (8.0) | 74.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 121 | 249
  Male | 84 | 101 | 185
Region of Enrollment [Number; unit: participants]
  China | 212 | 222 | 434

OUTCOME MEASURES:

1. Primary Outcome: Decision to Undergo Cataract Surgery (Surgery Acceptance)
Description: Measured as a percentage of subjects who decide to undergo cataract surgery within 6 months after screening (positive) out of total subjects.
Time Frame: within 6 months after screening examination
Population: All participants who completed the study were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of participants | 31.1 | 34.2

2. Secondary Outcome: Attendance at Hospital for Pre-operative Examination
Description: Measured as a percentage of people who presented to the hospital within 6 months after screening (positive) out of total subjects.
Time Frame: within 6 months after screening examination
Population: All participants who completed the study were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of participants | 40.1 | 41.4

3. Secondary Outcome: Knowledge That Cataract Can be Treated
Description: Measured as a percentage of subjects who correctly answer the question in a questionnaire.
Time Frame: Assessed during day of screening examination
Population: Analysis was conducted for all participants who responded to this question in the survey.
Measure: Number; unit: percentage of respondents
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of respondents | 87.7 | 79.7

4. Secondary Outcome: Belief That Surgery Will be Painful
Description: Measured as a percentage of subjects who agree with the statement in a questionnaire.
Time Frame: Assessed during day of screening examination
Population: Analysis was conducted for all participants who responded to this question in the survey.
Measure: Number; unit: percentage of respondents
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of respondents | 48.1 | 57.7

5. Secondary Outcome: Belief That Vision Will Improve "a Lot" Following Surgery
Description: Measured as a percentage of subjects who agree with the statement in a questionnaire.
Time Frame: Assessed during day of screening examination
Population: Analysis was conducted for all participants who responded to this question in the survey.
Measure: Number; unit: percentage of respondents
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of respondents | 62.0 | 54.0

6. Secondary Outcome: Belief That Surgeons at the Hospital Are "Highly Skilled"
Description: Measured as a percentage of subjects who agree with the statement in a questionnaire.
Time Frame: Assessed during day of screening examination
Population: Analysis was conducted for all participants who responded to this question in the survey.
Measure: Number; unit: percentage of respondents
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of respondents | 74.1 | 79.4

7. Secondary Outcome: Belief That Doctors and Nurses at the Hospital Have "Very Good" Attitudes
Description: Measured as a percentage of subjects who agree with the statement in a questionnaire.
Time Frame: Assessed during day of screening examination
Population: Analysis was conducted for all participants who responded to this question in the survey.
Measure: Number; unit: percentage of respondents
Arm/Group | Counseling | Non-counseling
Number analyzed (Participants) | 212 | 222
percentage of respondents | 81.9 | 82.9

ADVERSE EVENTS:
Arm/Group | Counseling | Non-counseling
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/222
Other Adverse Events (participants affected / at risk) | 0/212 | 0/222

LIMITATIONS AND CAVEATS:
One of the six participating hospitals did not adhere to protocol, and thus total number of subjects analyzed was smaller than originally anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes